CLINICAL TRIAL: NCT00285948
Title: Primary Birmingham Hip Resurfacing Arthroplasty Using a Metal-on-Metal Couple in the Young Active Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: René Verdonk, University Hospital Ghent
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004/339
Record Dates: First submitted 2006-02-01; First posted 2006-02-02 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Indications for a Total Hip Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Primary Birmingham hip resurfacing arthroplasty using a metal-on-metal couple

SUMMARY:
To prospectively obtain data about the clinical and radiological results of the resurfacing technique as primary hip prosthesis in young active patients

ELIGIBILITY:
Inclusion Criteria:

* Total hip prosthesis

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 1998-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Clinical and radiological results

CONTACTS AND LOCATIONS:
Overall Officials: Rene Verdonk, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be